CLINICAL TRIAL: NCT06968637
Title: Improving Patient-centered Care for Diabetes in Bangladesh Through "Dynamic Integration" of Vision Care on the Supply Side
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orbis (Other)
Collaborators: District Diabetes Hospital, Dinajpur district of Bangladesh (Unknown); Gausul Azam BNSB Eye Hospital in the Dinajpur district of Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PIS-DR-SUPPLY-2025
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy (DR)
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Cluster-randomised design, with diabetologist as the cluster. In the intervention group, a Patient Information System (PIS) database will be used, both at the diabetic hospital and eye hospital in Dinajpur. The PIS will be used for referral tracking, to deliver the results of the eye exam to the diabetologist, and, most importantly, based on the result of the DR exam, to provide specific care recommendations for diabetes management. Based on existing guidelines, when DR is present, the PIS will prompt diabetologists to check, and if necessary, change medicines to optimize, blood sugar, blood pressure and lipids. Therefore, through the doctors of the diabetic hospital tracking eye results, the PIS will reinforce the need for the patient to visit both the eye hospital and diabetic hospital for DM/DR management and will improve overall DM care.
  In the Control group, information on the DR exam will be conveyed through the PIS without specific care recommendations.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Only DR results provided (No Intervention): For these participants, the patient information system (PIS) will send only diabetic retinopathy (DR) results to the Diabetologist at the diabetic hospital without specific care recommendations
- Intervention Group: DR results + care recommendations for DM management provided (Experimental): For these participants, the patient information system (PIS) will send DR results to the Diabetologist at the diabetic hospital along with specific care recommendations for diabetes management (only for those patients with ANY DR)
  Interventions: Other: care recommendations

INTERVENTIONS:
Other: care recommendations — Provision of specific care recommendations for diabetes management. Based on existing guidelines, when any DR is present, the PIS will prompt diabetologists to check, and if necessary, change medicines to optimize, blood sugar, blood pressure and lipids.
  Other Names: Specific DM care recommendations
  Arms: Intervention Group: DR results + care recommendations for DM management provided

SUMMARY:
The goal of this clinical trial is to determine whether integration of vision care into the DM treatment system, by providing specific recommendations to doctors for management of diabetes alongside feedback on positive eye exams for DR can improve diabetes care outcomes.

The main questions it aims to answer are:

1. Does delivery of specific diabetes management recommendations to diabetes doctors for patients of theirs found to have DR lead to significantly improved blood glucose control as indicated by % reaching WHO targets of HbA1c (or targets for blood sugar if HbA1c data are unavailable)?
2. What is the cost-effectiveness of the intervention, measured as total intervention cost per additional participant reaching the WHO target?

Researchers will compare participant adherence with international guidelines when DR results are provided by a PIS without specific care recommendations to when the PIS provides DR results with specific care recommendations for DM management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DM
* Diagnosed with DR in at least one eye
* Over 30 years of age
* Currently treated at the Dinajpur Diabetes Hospital and Gausul Azam BNSB Eye Hospital in Bangladesh
* willingness to participate in the study

Exclusion Criteria:

* Any ocular condition impairing the view of the fundus sufficiently to preclude grading of the image for DR.
* Inability to comply with retinal photography to the extent that a gradable image cannot be captured, or any other factor leading to absence of sufficient images to grade at least one eye of a participant.
* Medical conditions that could impair compliance with follow-up (such as stroke, dementia, etc.)
* Unwilling to participate in the study, or incapable of giving informed consent.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants reaching WHO target HbA1c levels of <= 7.0% (or WHO blood sugar targets if HbA1c data are unavailable) among participants with any DR, upon chart review by a masked clinician observer, compared between study groups. | From enrollment to chart review (3 months after enrollment)
  According to the World Health Organization (WHO), the specific HgA1c target is <= 7.0%

SECONDARY OUTCOMES:
Cost-effectiveness, measured as total intervention cost per additional patient meeting the WHO blood sugar target. | Enrollment to chart review (3 months after enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Munir Ahmed, Principal Investigator — Orbis Bangladesh; Nathan Congdon, Principal Investigator — Orbis
Locations (2):
- Bangladesh (2):
  - Dinajpur Diabetes & Swasthoseba Hospital, Dinajpur Sadar, Dinajpur
  - Gausul Azam BNSB Eye Hospital, Dinajpur District

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be shared upon reasonable request to the corresponding author
Supporting Information: Study Protocol, SAP, ICF